CLINICAL TRIAL: NCT05392036
Title: : Effects of Therapeutic Ultrasound Versus Shockwave Therapy on Pain, Range of Motion and Function in Recreational Runners With Medial Tibial Stress Syndrome
Brief Title: Effects of Therapeutic Ultrasound Versus Shockwave Therapy in Medial Tibial Stress Syndrome in Recreational Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0139 Khizra
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Medial Tibial Stress Syndrome
Keywords: Shock wave; medial tibial stress syndrome; Ultrasound
MeSH Terms: conditions — Medial Tibial Stress Syndrome | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): shockwave therapy
  Interventions: Other: baseline physical therapy treatment along with shockwave therapy
- Group B (Other): therapeutic ultrasound
  Interventions: Other: baseline physical therapy treatment along with therapeutic ultrasound

INTERVENTIONS:
Other: baseline physical therapy treatment along with shockwave therapy — Group A, this group will receive conventional therapies along with shockwave therapy. Basic treatment includes icing (15-20 min) to control inflammation, rest, cessation of pain causing activity, anti-inflammatory (NSAIDs) and basic stretching and strengthening exercises. Shockwave therapy is a non-invasive therapeutic modality with convenience, effectiveness and safety. It is used to treat various musculoskeletal disorders without surgery. A session of 30-45 min will include icing 15 min and 5-10 min of shock wave therapy session will be commenced with strengthening and stretching exercises.
  Arms: Group A
Other: baseline physical therapy treatment along with therapeutic ultrasound — This group will receive therapeutic ultrasound along with conventional treatment. Conventional therapy includes icing, rest, anti-inflammatory drugs, and basic strengthening and stretching exercises. A session of 30-45 min will include icing for 10-15 min therapeutic ultrasound 15min with a frequency 1-3MHz and the session will be ended with strengthening and stretching exercises.
  Only eligible patients who have fulfilled the inclusion criteria will be included. A daily session of 30-45min for 2 consecutive weeks will be given. A baseline assessment will be done and the patient will be allocated randomly to both groups for two weeks. Re-assessment will be done after 2 weeks. For long term, effects re-assessment will be done after 6 weeks
  Arms: Group B

SUMMARY:
This project was a Randomized control trial conducted to check the effects of therapeutic ultrasound versus shockwave therapy on pain , range of motion and function in recreational runners with medial tibial stress syndrome so that we can formulate a better and most effective regime for treatment of medial tibial stress. Duration was of 6 months, convenient sampling was done, subject following eligibility criteria from Ghurki Trust teaching hospital, horizon hospital and surgimed hospital. Group A participants were given baseline treatment along with shockwave and Group B were given baseline treatment along with therapeutic ultrasound. Assesment was done at baseline and at 2nd week and 6th week post-interrvention . Assessment was done via, Numeric pain rating scale(NPRS), Lower Extermity functional scale LEFS ) and goniometric measurements of shoulder ranges, data was analyzed by using SPSS version 26.

DETAILED DESCRIPTION:
Medial tibial stress syndrome (MTSS) is a common low leg injury. It is described as activity-induced pain along posterior medial border of leg approximately for 5 cm. Most commonly reported by runners and military personnel. Incidence of MTSS ranges between 13.6% to 20% in runners. Significant increase in loading activities or rigorous exercise causing high impact like skiping, jogging can induce MTSS which leads to stress fracture of tibia. Various risk factors are associated with the incidence of medial tibial stress syndrome which includes both intrinsic and extrinsic factors. Current study has involved comparison of therapeutic ultrasound versus shockwave therapy as there is limited knowledge about comparison of therapeutic ultrasound versus shockwave therapy.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Pain at distal 2/3 of tibia
* Previous history of MTSS
* Recreational runner

Exclusion Criteria:

* History of lower limb fracture

  * Any lower limb surgical history
  * Any malignancy
  * Professional athlete
  * Cardiopulmonary insufficiency

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
LEFS | 3rd day
  It is used to assessment of lower extremity function a questionnaire of 20 questions about a person also ability to perform daily task 0 is minimum score, 80 is maximum score. lower the score greater the disability.
Goniometry | 3rd day
  A goniometer is an instrument which measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Ghurki Trust Hospital, Horizon Hospital, Surgimed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McClure CJ, Oh R. Medial Tibial Stress Syndrome. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538479/ PMID 30860714
- [Background] Okunuki T, Koshino Y, Yamanaka M, Tsutsumi K, Igarashi M, Samukawa M, Saitoh H, Tohyama H. Forefoot and hindfoot kinematics in subjects with medial tibial stress syndrome during walking and running. J Orthop Res. 2019 Apr;37(4):927-932. doi: 10.1002/jor.24223. Epub 2019 Feb 12. PMID 30648281
- [Background] Menendez C, Batalla L, Prieto A, Rodriguez MA, Crespo I, Olmedillas H. Medial Tibial Stress Syndrome in Novice and Recreational Runners: A Systematic Review. Int J Environ Res Public Health. 2020 Oct 13;17(20):7457. doi: 10.3390/ijerph17207457. PMID 33066291
- [Background] Wang CJ. Extracorporeal shockwave therapy in musculoskeletal disorders. J Orthop Surg Res. 2012 Mar 20;7:11. doi: 10.1186/1749-799X-7-11. PMID 22433113
- [Background] Tsai WC, Tang ST, Liang FC. Effect of therapeutic ultrasound on tendons. Am J Phys Med Rehabil. 2011 Dec;90(12):1068-73. doi: 10.1097/PHM.0b013e31821a70be. PMID 21552108
- [Background] Gomez Garcia S, Ramon Rona S, Gomez Tinoco MC, Benet Rodriguez M, Chaustre Ruiz DM, Cardenas Letrado FP, Lopez-Illescas Ruiz A, Alarcon Garcia JM. Shockwave treatment for medial tibial stress syndrome in military cadets: A single-blind randomized controlled trial. Int J Surg. 2017 Oct;46:102-109. doi: 10.1016/j.ijsu.2017.08.584. Epub 2017 Sep 5. PMID 28882773
- [Background] Naderi A, Bagheri S, Ramazanian Ahoor F, Moen MH, Degens H. Foot Orthoses Enhance the Effectiveness of Exercise, Shockwave, and Ice Therapy in the Management of Medial Tibial Stress Syndrome. Clin J Sport Med. 2022 May 1;32(3):e251-e260. doi: 10.1097/JSM.0000000000000926. Epub 2021 Mar 24. PMID 33797477
- [Background] Moen MH, Holtslag L, Bakker E, Barten C, Weir A, Tol JL, Backx F. The treatment of medial tibial stress syndrome in athletes; a randomized clinical trial. Sports Med Arthrosc Rehabil Ther Technol. 2012 Mar 30;4:12. doi: 10.1186/1758-2555-4-12. PMID 22464032
- [Background] Mendez-Rebolledo G, Figueroa-Ureta R, Moya-Mura F, Guzman-Munoz E, Ramirez-Campillo R, Lloyd RS. The Protective Effect of Neuromuscular Training on the Medial Tibial Stress Syndrome in Youth Female Track-and-Field Athletes: A Clinical Trial and Cohort Study. J Sport Rehabil. 2021 Apr 20;30(7):1019-1027. doi: 10.1123/jsr.2020-0376. PMID 33883301
- [Background] Yamasaki S. A Review of the Treatment and Prevention Options for Medial Tibial Stress Syndrome. 2019.